CLINICAL TRIAL: NCT01504893
Title: Multicenter Randomized Trial on Protective Ventilation Versus Conventional Ventilation During OLV in Patients Undergoing Thoracic Surgery
Brief Title: Very Low Tidal Volume vs Conventional Ventilatory Strategy for One-lung Ventilation in Thoracic Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera S. Maria della Misericordia (Other)
Responsible Party: Principal Investigator, Giorgio Della Rocca, M.D., Azienda Ospedaliera S. Maria della Misericordia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ALI01
Record Dates: First submitted 2011-12-30; First posted 2012-01-06 (Estimated); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: One lung ventilation; PEEP; thoracic surgery; lobectomy and pneumonectomy; ARDS
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Protective (Experimental): Two-lung ventilation (TLV): tidal volume = 8 mL / kg PBW, peak airway pressure ≤ 25 cm H2O, I: E = 1:2; after lung re-expansion to the closure of the chest will set a PEEP of 5 cmH2O
  OLV (OLV): 4 mL / kg PBW, peak airway pressure ≤ 35 cmH2O, respiratory rate <30, I:E = 1:2 / 1:3.
  During OLV in case of desaturation (before increasing the FiO2) and every 60 minutes alveolar recruitment maneuvers followed by the setting of PEEP to 5 cmH2O
  Interventions: Procedure: Protective one lung ventilation
- Conventional (No Intervention): Two-lung ventilation (TLV): tidal volume = 8 mL / kg PBW, peak airway pressure ≤ 25 cmH2O; I: E = 1:2; after lung re-expansion to the closure of the chest PEEP set to 5 cmH2O
  OLV (OLV): 6 mL / kg PBW, peak airway pressure ≤ 35 cmH2O; I: E = 1:2.

INTERVENTIONS:
Procedure: Protective one lung ventilation — Low tidal volume, PEEP and alveolar recruitment maneuver
  Arms: Protective

SUMMARY:
The purpose of this study is to determine if a protective ventilatory strategy during one-lung ventilation (OLV) based on low tidal volume, PEEP and alveolar recruitment maneuver can reduce Acute Respiratory Distress Syndrome (ARDS) and Postoperative pulmonary complications (PPCs) after major pulmonary resection.

Primary endpoint: Evaluation of postoperative ARDS incidence

Secondary endpoint: Evaluation od PPC incidence and postoperative outcomes (other complications, unplanned Intensive Care Admission, hospital and ICU length of stay, in-hospital mortality)

DETAILED DESCRIPTION:
Pulmonary postoperative complications (PPCs) are the most frequent adverse events after thoracic surgery. Acute respiratory distress syndrome (ARDS) is the most severe among PPCs. Injurious mechanical ventilation is a recognized risk factor associated with ARDS and PPCs after major thoracic surgery.

International literature reports a wide use of tidal volume around 5-6 ml/kg predicted body weight (PBW) during one lung ventilation (OLV) but variable use of PEEP and alveolar recruitment maneuver (ARM).

The aim of this multicenter, randomized, single blind study is to determine if a protective ventilatory strategy during OLV based on low tidal volume, PEEP and alveolar recruitment maneuver compared to conventional strategy can reduce ARDS and PPCs after major pulmonary resection.

Primary outcome is the incidence of in-hospital ARDS.

Secondary outcomes are in-hospital incidence of postoperative pulmonary complications (PPCs), major cardiovascular events, unplanned Intensive Care Unit admission, in-hospital length of stay and mortality

RANDOMIZATION

Patients are randomly assigned to receive protective or conventional OLV according to a computer-generated randomization list (1:1 ratio) before anesthesia induction.

Patients are blinded to the treatment. Anesthesiologists and surgeons are unblinded to the treatment during the surgical procedure and the postoperative outcome assessment.

MEASUREMENTS

Intraoperative collection of ventilatory settings, airway pressures, arterial blood gases analysis at the following time points:

T1: two lung ventilation in supine position before placing the patient in lateral decubitus; T2: 30 minutes after OLV start; T3: 60 minutes after OLV start; T4: 20 minutes after lobectomy/pneumonectomy (during OLV); T5: 15 minutes after ARM in supine position and during two lung ventilation.

Postoperative data collection 1, 12, 24, 36, 48 hours after surgery and at discharge. Arterial blood gas analysis will be performed 1 hour after extubation and 24 and 72 hours after surgery (or in case of respiratory insufficiency).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years
* ASA IV
* Elective thoracotomies or thoracoscopic major lung resection surgery (lobectomy, bilobectomy, pneumonectomy)

Exclusion Criteria:

* Emergency surgery
* Wedge resection or atypical resection
* Non-resective lung surgery requiring OLV
* Patients < 18 years
* BMI < 20 and BMI > 29
* Heart disease with ejection fraction <50% and/or severe valvulopathy
* Pulmonary hypertension
* Renal failure requiring dialytic treatment
* Drug addiction
* Mental retardation, depression and psychiatric disease
* Motor or sensory deficit
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 984 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Acute Respiratory Distress Syndrome (ARDS) incidence | Hospital stay (7 days average expected)
  incidence of ARDS (%)

SECONDARY OUTCOMES:
Postoperative pulmonary complications (PPCs) | Hospital stay (7 days average expected)
  Incidence of PPCs (%)
In-hospital mortality | Hospital stay (7 days average aspected)
  To determine mortality (%)
Postoperative complications | Hospital stay (7 days average expected)
  To determine how many patients (%) would have any postoperative complications
Unplanned Intensive Care Unit (ICU) admission | Hospital stay (7 days average aspected)
  To determine how many patients would require an ICU admission (%)
Intensive Care Unit (ICU) Length of stay | Hospital stay (7 days average aspected)
  Length of stay in ICU (days)
Length of hospital stay | Hospital stay (7 days average expected)
  Duration of hospital length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Della Rocca, MD, Prof, Principal Investigator — Azienda Ospedaliero-Universitaria S. Maria della Misericordia - Udine. Italy
Locations (16):
- Italy (16):
  - ASST Papa Giovanni XXIII, Bergamo
  - IRCCS Policlinico Sant'Orsola-Malpighi, Bologna
  - Ospedale Centrale, Bolzano
  - Azienda Ospedaliera Brotzu - Ospedale Oncologico Businco, Cagliari
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Fondazione IRCCS Istituto Nazionale Tumori, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Azienda Ospedaliera-Universitaria, Modena
  - Istituto Nazionale Tumori Fondazione Pascale, Napoli
  - Azienda Ospedaliero-Universitaria, Padua
  - IRCCS Centro di Riferimento Oncologico della Basilicata, Rionero in Vulture
  - Istituto Nazionale Tumori Regina Elena, Rome
  - Azienda Ospedaliera Universitaria Senese, Siena
  - Ospedale di Cattinara, Trieste
  - Department of Anesthesia and Intensive Care Unit, Udine
  - Ospedale di Circolo e Fondazione Macchi, Varese

REFERENCES:
- [Background] Yang M, Ahn HJ, Kim K, Kim JA, Yi CA, Kim MJ, Kim HJ. Does a protective ventilation strategy reduce the risk of pulmonary complications after lung cancer surgery?: a randomized controlled trial. Chest. 2011 Mar;139(3):530-537. doi: 10.1378/chest.09-2293. Epub 2010 Sep 9. PMID 20829341
- [Background] Licker M, Diaper J, Villiger Y, Spiliopoulos A, Licker V, Robert J, Tschopp JM. Impact of intraoperative lung-protective interventions in patients undergoing lung cancer surgery. Crit Care. 2009;13(2):R41. doi: 10.1186/cc7762. Epub 2009 Mar 24. PMID 19317902